CLINICAL TRIAL: NCT05962723
Title: Pancreatic Cyst Fluid Glucose: New Armamentarium in the Diagnosis of Mucinous Pancreatic Cystic Lesion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: Pancreatic cyst glucose 1; NCT06189339 (obsolete NCT alias)
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Cyst Fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — cystic fluid glucose level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: EUS — EUS examination and cystic fluid will be aspirated for analysis, including cystic fluid Glucose, CEA, amylase. Morey's biopsy will be done in the cases feasible for biopsy.

SUMMARY:
All participants undergoing radiological imaging and found to have pancreatic cyst of size > 2cm will be subjected to EUS (Endoscopic ultrasound) examination and cystic fluid will be aspirated for analysis, including cystic fluid Glucose, CEA, amylase. Morey's biopsy will be done in the cases feasible for biopsy. The sensitivity and specificity of cystic fluid glucose level will be analysed taking CEA (carcinoembryonic antigen) level with EUS findings, amylase level as gold standard for diagnosis, in cases with no surgical management.

DETAILED DESCRIPTION:
Pancreatic cystic lesion prevalence noted to be increased dramatically in last few decades. Earlier record showed the prevalence rate of 2.4-2.6% with magnetic resonance imaging (MRI), though sometimes reaching 13.5%.Recent study showed prevalence of pancreatic cysts to be 49%. Most of the pancreatic cyst are benign and require conservative management and regular evaluation only. Malignant cystic lesion on the other hand require immediate attention and surgical excision in most of cases. Thus, diagnosis of pre-malignant & malignant pancreatic cyst are essential, to predict the prognosis and decide further management.

Most widely accepted biochemical test for preoperative differentiation of mucinous from benign pancreatic cysts is cystic fluid carcinoembryonic antigen (CEA). CEA with cutoff value of 192 ng/ml has sensitivity, specifivcity and accuracy of 75%, 84% & 79% respectively. This is expensive and requires a longer duration for obtaining the results. Few recent studies proposed the role of cystic fluid glucose level in the diagnosis of malignant cyst.

ELIGIBILITY:
Inclusion Criteria:

* Patients (between 18 to 60 years of age)
* Pancreatic cyst of size >2 cm noted on radiological imaging

Exclusion Criteria:

* Patient's age <16yrs or >80 yrs.
* Prior history of pancreatitis (within 3 months)
* Pregnant female
* Unfit for endoscopic ultrasound
* Not wiling for consent

Ages: 18 Minutes to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with pancreatic cyst of size >2 cm, seen on radiological image, having no contraindication for endoscopic ultrasound and has not suffered from pancreatitis within last 3 months) coming to OPD/admitted in ward in AIG Hospital , Hyderabad satisfying inclusion and exclusion criteria after informed consent, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity and accuracy | One Year
  sensitivity, specificity and accuracy of pancreatic cystic fluid glucose level with comparison to fluid CEA levels, morey's biopsy result and surgical findings.

IPD SHARING:
Plan to Share IPD: No